CLINICAL TRIAL: NCT02508727
Title: Myocardial Deformation in Real-time 3D Ultrasound. Normal Values in Adults and Validation Against the Tagged MRI
Acronym: DIRECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 10-156
Record Dates: First submitted 2015-07-23; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Healthy volunteers (Other): Healthy volunteers
  Interventions: Other: MRI; Other: 3D cardiac ultrasound
- Subjects with an anterior myocardial infarction sequela (Other): Subjects with an anterior myocardial infarction sequela
  Interventions: Other: MRI; Other: 3D cardiac ultrasound
- Subjects with lower myocardial infarction sequelae (Other): Subjects with lower myocardial infarction sequelae
  Interventions: Other: MRI; Other: 3D cardiac ultrasound

INTERVENTIONS:
Other: MRI
Other: 3D cardiac ultrasound

SUMMARY:
Cardiac exploration almost systematically requires the acquisition and / or calculating function indices. The ejection fraction (LVEF) is probably based index most widely used in all cardiac exploration methods. This relatively universal overall index has very many qualities. LVEF is widely used in clinical practice through the exploration and monitoring of all heart disease.

Current progress in the management of various cardiomyopathies pass through the detection of early attacks. This testing often takes place upstream changes in LVEF that remains long normal or normalized. Sensitive indicators capable of detecting early abnormalities of regional functions are essential in addition to conventional echocardiography. Various studies have shown the contribution of these new markers in early detection of abnormalities of the cardiac function. The most widely used indicator in these studies because of its high sensitivity to analyze the movements of the heart is the tissue Doppler. Tissue Doppler however has limitations in particular its dependence on the incident angle, which makes it impossible to correct analysis of non-aligned in the axis of the ultrasonic beam components.

A new way of exploring the regional function of the heart, speckle tracking, can analyze heart deformations along the principal axes of the heart. The advantage of this technique has been shown in various pathological situations. Currently, this technique is mostly used in longitudinal and transverse view 2D imposing multiple planes cuts. 3D potential of this technique is not currently known, acquisition of 3D technology is recent (2004) and dedicated software is confidential dissemination and unvalidated.

The validated technique, 3D reference analysis of myocardial deformation is tagged MRI. In the 90s, studies have demonstrated the feasibility of this technique, the ability to access all of the myocardial deformation in space and to define normal values. The cost of the procedure, duration, limited accessibility and post-processing very time consuming limited the scope of the clinical benefits of this modality.

Echocardiography has major advantages over MRI, particularly its high availability, low cost and flexibility of use. The ability to access with MRI as the 3D deformation of the heart is a new opportunity that it is essential to validate.

The main purpose of the study is to compare the strain values obtained 3D ultrasound to those obtained by MRI tagged in a control group and a group of subjects with an anterior infarction sequela.

ELIGIBILITY:
Inclusion Criteria:

* Patients who signed the consent form
* Beneficiaries of the health security system
* No known cardiovascular disease to healthy subjects or patient having a previous heart attack or less proved by cardiac MRI or viability of myocardial scintigraphy performed before. The infarct zone is defined as the area of delayed enhancement cardiac MRI signal in 10-15 minutes after gadolinium injection.

Exclusion Criteria:

* Age <18 years
* Adult guardianship
* Contraindications to MRI: metallic implants, pacemaker, implantable defibrillator, claustrophobia
* For patients only: Contraindication to Dotarem (renal failure with creatinine clearance <30 ml / min / 1.73m2 according to MDRD formula, known allergy to gadolinium salts)
* Pregnant and or lactating
* Recent acute coronary syndrome (<6 weeks)
* Ventricular arrhythmias and supra ventricular significant
* Heart failure stage III-IV NYHA
* Unbalanced severe hypertension (BP> 160/110 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Strain value | baseline
  Comparison beetween arms and taage MRI and 3D cardiac echography

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, Basse Normandie, France